CLINICAL TRIAL: NCT06545630
Title: Tumor Antigen-sensitized DC Vaccine as an Adjuvant Therapy for R0 Resection of Colorectal Cancer Liver Metastases
Brief Title: Tumor Antigen-sensitized DC Vaccine for Colorectal Cancer Liver Metastases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Meng Qiu, Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeoDC-CRC-01
Record Dates: First submitted 2024-07-01; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-07

CONDITIONS: Carcinoma; Colorectal Cancer
MeSH Terms: conditions — Carcinoma; Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant Group/Arm (Experimental): Tumor antigen-sensitized vaccine is administrated, 1-week interval, totally 2 times.
  2-week later, Neo-antigen DC vaccine is administrated, 2-week interval, totally 5 times.
  According to the conditions of patients, it will be used for five more times
  Interventions: Biological: Tumor antigen-sensitized DC vaccine

INTERVENTIONS:
Biological: Tumor antigen-sensitized DC vaccine — subcutaneous administration

SUMMARY:
The aim of this study is to explore the safety and efficacy of tumor antigen-sensitized DC vaccine in postoperative adjuvant treatment of R0 excision Colorectal Cancer Liver Metastases.

ELIGIBILITY:
Inclusion Criteria:

Pathologically confirmed diagnosis of colorectal cancer； Karnofsky performance status 0-1; Patients with tumors identified by pathologic immunohistochemistry as pMMR or by genetic testing as MSS/MSI-L; Imaging diagnosis of stage IV, resection of both primary and metastatic tumors and had NED status after surgery; With a high risk of recurrence, such as liver metastasis CRS score >3 or successful conversion therapy; Multiple peritoneal metastases after CC0; Function of the main organs is normal; Edition Patient's written informed consent

Exclusion Criteria:

Tumor emergencies; Abnormal coagulation function; Contagious diseases, such as HIV, HBV, HCV infection; Mental disorders; Concomitant tumors; Immunological co-morbidities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival | Up to 18 months
  Time from assignment to treatment arm until a recurrence or progression of the disease

SECONDARY OUTCOMES:
Adverse Events Related to Treatment | Up to 12 months
  Rate of Adverse Events (AEs) related to the niraparib and dostarlimab combination per CTCAE v5.0
Overall Survival (OS) | Up to 36 months
  Time from assignment to treatment arm until death due to any cause
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 month after the last administration of Tumor Antigen-sensitized DC Vaccine
  Adverse events (AE) will be graded and documented according to NCI-CTC AE v4.0 from the beginning of treatment to 1 months after the last date of treatment. Documentary will include severity, lasting period and occurrence time. Main AEs include hypertension, albuminuria, skin reaction of hands and feet, hemorrhage, dysphonia, transaminase rise, abdominal pain / abdominal discomfort, blood bilirubin rise, thyroid dysfunction, infection, diarrhea, fatigue / fatigue, appetite decline, oral mucositis, weight loss, fecal occult blood and platelet count decline

CONTACTS AND LOCATIONS:
Locations (1):
- Colorectal Cancer Center, West China Hospital, Chengdu, Chengdu/Sichuan, China

IPD SHARING:
Plan to Share IPD: No